CLINICAL TRIAL: NCT03941470
Title: Assessment of Natural Killer Cells Activating and Inhibitors
Brief Title: Assessment of Natural Killer Cells in Unexplained Recurrent Pregnancy Loss
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yossra Mahmoud Mohammed, Assesment of Natu, Assiut University
Other Study IDs: 17200339
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Female; Recurrent Miscarriage; Unexplained Pregnancy Loss
Keywords: NK ;natural killer cells
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- unexplained recurrent pregnancy loss: peripheral blood sample examined by flowcytometry
- control fertile multipara: peripheral blood sample examined by flowcytometry

SUMMARY:
To assess natural killer cells frequency and activation in cases of unexplained recurrent abortion in comparison to fertile cases

* 2. . To study the expression of stimulatory receptors of natural killer cell.
* 3-To study the expression of inhibitory receptors of natural killer cell.

DETAILED DESCRIPTION:
NK-cell functioning is controlled by a wide range of receptors that are expressed on the cell surface. These receptors are either inhibitory or activating in nature. The family of inhibitory receptors consists of the killer immunoglobulin-like receptors (KIR) or Ig-like receptors (CD158), the C type lectin receptors (CD94-NKG2A) and leukocyte inhibitory receptors (LIR1, LAIR-1). Activating receptors are the natural cytotoxic receptors (NKp46, NKp44), C type lectin receptors (NKG2D, CD94-NKG2C), and Ig-like receptors (2B4). A particular NK cell typically expresses two to four inhibitory receptors in addition to an array of activation receptors. The killing by NK cells is mediated through several activating NK receptors. Among these are NKG2D and the three natural cytotoxicity receptors (NCRs), NKp30, NKp44, and NKp46 (Yang et al., 2000) Osne of the natural cytotoxicity receptors (NCRs) NKp46, , is a unique marker that functions in NK cell cytotoxicity and cytokine production. Expression of NKp46 on NK cells is lower in women with recurrent pregnancy loss, so evaluation of NKp46 on peripheral blood NK cells may provide a means of screening for reproductive abnormalities (Fukui et al., 2015).

During pregnancy, decidual NK cells comprise ∼70-80% of the decidual lymphocytes and are considered a special NK subset that does not exert cytolytic functions against trophoblast cells and has generally reduced cytotoxicity (Hanna and Mandelboim, 2007).

These cells express activating NK receptors, including all the NCRs and NKG2D. However, instead of triggering cytotoxicity, these receptors act to stimulate secretion of cytokines and angiogenic factors, which are essential for trophoblast invasion and vascular modifications (Hanna et al., 2006).

One study reported that pNK cell levels show changes in decidual NK cell levels (Park et al., 2010). Whereas some other reports have shown that the assessment of peripheral blood NK cells would not

ELIGIBILITY:
Inclusion Criteria:

* 1.Age less than 40 years. 2.History of two or more spontaneous miscarriages .

Exclusion Criteria:

* 1. Age more than 35 years. 2. Women with elevated level of TSH above (2.5 mIU/ml) or prolactin above( 19.5 ng/mL)and uncontrolled DM.

  3. Women with autoimmune disorder (antiphospholipid antibody syndrome)with LA1/LA2 ratio more than( 1.2).

  4.Women receiving oral contraceptive pills.

Max Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We will recruit patients from outpatient clinics from Assuit University Hospital,Women fulfilling eligibility criteria will be included after careful gynecologycal examination,Those who consent to participate will be referred to the lab for investigation.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-07-20 (Estimated)

PRIMARY OUTCOMES:
asses the number of Natural killer cells | 15 month
  flowcytometry

CONTACTS AND LOCATIONS:
Overall Officials: assiut university, Principal Investigator — Assiut University
Locations (1):
- Yossra Mahmoud Mohammed, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fukui A, Kamoi M, Funamizu A, Fuchinoue K, Chiba H, Yokota M, Fukuhara R, Mizunuma H. NK cell abnormality and its treatment in women with reproductive failures such as recurrent pregnancy loss, implantation failures, preeclampsia, and pelvic endometriosis. Reprod Med Biol. 2015 Apr 11;14(4):151-157. doi: 10.1007/s12522-015-0207-7. eCollection 2015 Oct. PMID 29259412
- Available data/document: Study Protocol: IRB17200056 — http://Email:ethics_committee12@yahoo.com